CLINICAL TRIAL: NCT03881124
Title: Pain Trajectories in Severe Persistent Inguinal Post-herniorrhaphy Pain
Status: Completed | Type: Observational
Sponsor: University of Copenhagen (Other)
Responsible Party: Principal Investigator, mads u werner, Principal Investigator, University of Copenhagen
Other Study IDs: H-2-2011-023-TRJ
Record Dates: First submitted 2019-03-14; First posted 2019-03-19 (Actual); Last update posted 2024-02-22 (Actual); Status verified 2024-02

CONDITIONS: Chronic Pain
Keywords: Inguinal Herniorrhaphy; Hernia; Persistent postsurgical pain; Long term follow up; Quantitative sensory testing (QST); Pain trajectory; Explanatory variables
MeSH Terms: conditions — Chronic Pain; Hernia; Pain, Postoperative

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Severe persistent postsurgical pain (PPP) remains a major healthcare challenge. In the third most common surgical procedure in the UK, inguinal herniorrhaphy, including 85,000 surgeries in 2015, an estimated 1,500 to 3,000 patients will annually develop severe PPP. While the trajectory of PPP is generally considered a continuation of the acute post-surgery pain, recent data suggest the condition may develop with a delayed onset. The present study evaluated pain-trajectories in a consecutive cohort referred to a tertiary PPP-center. Explanatory variables based on individual psychometric, sensory and surgical profiles were analysed.

DETAILED DESCRIPTION:
Severe persistent post-surgical pain (PPP) is a prevalent medical problem leading to impairment of physical and psycho-social functions in a large number of individuals.Severe PPP may significantly influence 4-8% of the surgical population, depending primarily on the surgical procedure and technique, but also patient-related pre-surgical factors.Updated criteria for PPP have recently been suggested. Inguinal herniorrhaphy qualifies for PPP-research due to a high surgical volume. Paradoxically, while the surgery is considered a minor procedure with limited tissue damage it is carried out in a territory with abundant nerve and vascular supply, and, complex musculoskeletal functions essential for locomotor actions. Persistent pain after inguinal herniorrhaphy may develop after a seemingly successful surgical procedure, and, is seen in a severe form in 2-4% of the patients associated with significant deterioration of the health-related quality of life.

The transition process from acute to persistent pain may be more complex than previously assumed, making the study of temporal pain trajectories interesting. Based on clinical experience from a nationwide research center in PPP following inguinal herniorrhaphy, the authors decided first, to perform a prospective exploratory cohort study examining graphical pain charts by planimetrics, attempting to construct a valid statistical sub-classification of the trajectories. Secondly, the relationship between the sub-classification of the trajectories, and, potential explanatory variables, based on individual profiles of pain, psychometrics, quantitative sensory testing, and surgical procedures, were analysed, using principal component analysis and logistic regression models.

ELIGIBILITY:
Inclusion Criteria:

* Patients with severe persistent pain (>6 mo) after groin hernia repair referred to our center for PPP

Exclusion Criteria:

* Unable to cooperate with the sensory examinations

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with severe persistent pain after groin hernia repair with psychophysical disability referred to a dedicated tertiary center on a nationwide basis.
Sampling Method: Non-Probability Sample
Enrollment: 95 (Actual)
Dates: Start 2014-08-21 (Actual); Primary Completion 2016-11-10 (Actual); Study Completion 2016-11-10 (Actual)

PRIMARY OUTCOMES:
Group I pain trajectories | 2014-2016
  Trajectories are examined by area-under-curve using normalized pain intensities (numeric rating scale values 0-10 [y-axis]) and normalized time points (years [x-axis]) in patients with sustained severe where the acute post-surgical pain continued into persistent post-surgical pain (PPP) with unchanged high-intensity pain
Group II pain trajectories | 2014-2016
  Trajectories are examined by area-under-curve using normalized pain intensities (numeric rating scale values 0-10 [y-axis]) and normalized time points (years [x-axis]) in patients where the acute post-surgical pain decreased significantly to low-intensity levels, but pain recurred developing into high-intensity PPP
Group III pain trajectories | 2014-2016
  Trajectories are examined by area-under-curve using normalized pain intensities (numeric rating scale values 0-10 [y-axis]) and normalized time points (years [x-axis]) in patients where repeat-surgery precipitated high-intensity PPP
Group IV pain trajectories | 2014-2016
  Trajectories are examined by area-under-curve using normalized pain intensities (numeric rating scale values 0-10 [y-axis]) and normalized time points (years [x-axis]) in patients where pre-surgical high-intensity pain continued unchanged post-surgically.

SECONDARY OUTCOMES:
Pain intensity | 2014-2016
  Numeric Rating Scale (NRS; 0-10 units)
Activity of Daily Living (ADL) score | 2014-2016
  Activities Assessment Scale (AAS; 8 specified physical activities; 0-8 units each)
Assessments of Anxiety and Depression | 2014-2016
  Hospital Anxiety and Depression Scale (HADS; 14 items scale; 0-21 units)
Assessment of Pain Catastrophizing | 2014-2016
  Pain Catastrophizing Scale (PCS; 13 item scale; 0-65 units)
Quantitative sensory testing (QST) | 2014-2016
  Mechanical and thermal detection and pain thresholds
painDETECT | 2014-2016
  Neuropathic pain questionnaire (15 items scale; 0-38 points; 0-12 points = neuropathic pain unlikely; 13-18 = existence of neuropathic pain cannot unambigously be rejected;19-38 points = neuropathic pain likely)
S-LANSS | 2014-2016
  Neuropathic pain questionnaire (7 items; minimal cumulated score 0 points, maximum cumulated score 24 points; a score of 12 or more suggests pain of predominantly neuropathic origin)

IPD SHARING:
Plan to Share IPD: Yes
Data will be made available as a supplement to the published scientific article.
Supporting Information: Study Protocol, CSR
Time Frame: AUG-2020; 10 years
Access Criteria: Publicly available data

REFERENCES:
- [Background] Chapman CR, Vierck CJ. The Transition of Acute Postoperative Pain to Chronic Pain: An Integrative Overview of Research on Mechanisms. J Pain. 2017 Apr;18(4):359.e1-359.e38. doi: 10.1016/j.jpain.2016.11.004. Epub 2016 Nov 28. PMID 27908839
- [Background] Pogatzki-Zahn EM, Segelcke D, Schug SA. Postoperative pain-from mechanisms to treatment. Pain Rep. 2017 Mar 15;2(2):e588. doi: 10.1097/PR9.0000000000000588. eCollection 2017 Mar. PMID 29392204
- [Background] Kehlet H, Jensen TS, Woolf CJ. Persistent postsurgical pain: risk factors and prevention. Lancet. 2006 May 13;367(9522):1618-25. doi: 10.1016/S0140-6736(06)68700-X. PMID 16698416
- [Background] Werner MU, Bischoff JM. Persistent postsurgical pain: evidence from breast cancer surgery, groin hernia repair, and lung cancer surgery. Curr Top Behav Neurosci. 2014;20:3-29. doi: 10.1007/7854_2014_285. PMID 24523139
- [Background] Werner MU, Kongsgaard UE. I. Defining persistent post-surgical pain: is an update required? Br J Anaesth. 2014 Jul;113(1):1-4. doi: 10.1093/bja/aeu012. Epub 2014 Feb 18. No abstract available. PMID 24554546
- [Background] Werner MU. Management of persistent postsurgical inguinal pain. Langenbecks Arch Surg. 2014 Jun;399(5):559-69. doi: 10.1007/s00423-014-1211-9. Epub 2014 May 23. PMID 24849039
- [Background] Gartner R, Jensen MB, Nielsen J, Ewertz M, Kroman N, Kehlet H. Prevalence of and factors associated with persistent pain following breast cancer surgery. JAMA. 2009 Nov 11;302(18):1985-92. doi: 10.1001/jama.2009.1568. PMID 19903919
- [Background] Reinpold WM, Nehls J, Eggert A. Nerve management and chronic pain after open inguinal hernia repair: a prospective two phase study. Ann Surg. 2011 Jul;254(1):163-8. doi: 10.1097/SLA.0b013e31821d4a2d. PMID 21562403
- [Background] McCarthy M Jr, Jonasson O, Chang CH, Pickard AS, Giobbie-Hurder A, Gibbs J, Edelman P, Fitzgibbons R, Neumayer L. Assessment of patient functional status after surgery. J Am Coll Surg. 2005 Aug;201(2):171-8. doi: 10.1016/j.jamcollsurg.2005.03.035. PMID 16038812